CLINICAL TRIAL: NCT02337933
Title: Effect of Ursolic Acid Administration on Insulin Sensitivity and Metabolic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Manuel González Ortiz, Researcher Professor, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UA-MS
Record Dates: First submitted 2015-01-09; First posted 2015-01-14 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Metabolic Syndrome X
Keywords: Metabolic Syndrome; Central Obesity; Insulin Sensitivity; Ursolic Acid; Triterpenoid
MeSH Terms: conditions — Metabolic Syndrome; Obesity, Abdominal; Insulin Resistance | interventions — Ursolic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ursolic acid (Experimental): Ursolic acid capsules, 150 mg, once a day before breakfast during 12 weeks
  Interventions: Drug: Ursolic acid
- Placebo (Placebo Comparator): Calcined magnesia capsules, 150 mg, once a day before breakfast during 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ursolic acid — Ursolic acid capsules of 150 mg extracted from rosemary, once a day before breakfast
  Other Names: Urson; Prunol; Micromerol; Malol
  Arms: Ursolic acid
Drug: Placebo — Calcined magnesia capsules of 150 mg, once a day before breakfast
  Other Names: Calcined magnesia
  Arms: Placebo

SUMMARY:
The metabolic syndrome is characterized by the presence of overweight/obesity, insulin resistance, hyperglycemia, dyslipidaemia and hypertension and an inflammatory state, which together increase the risk of developing cardiovascular disease (CVD) or diabetes mellitus type 2 (DM2). It is also characterized by a decreased insulin sensitivity, namely, lower ability of insulin to metabolize glucose, key in the physiopathogeny of disease process.

In the search for a pharmacological agent that can attend more components of the metabolic syndrome and above all improve insulin sensitivity to effectively prevent the development of CVD and DM2, ursolic acid is a promising compound.

Ursolic acid is a pentacyclic carboxylic acid present in medicinal herbs, parts of some fruits like apple peel, and plants such as rosemary. There is scientific evidence of important benefits of ursolic acid level in vitro and in vivo on insulin, metabolism of lipids and glucose, as well as on the body weight and metabolic parameters. However, the results are not clear and the mechanisms are not fully elucidate.

The aim of this study is to evaluate the effect of ursolic acid on the insulin sensitivity and metabolic syndrome.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trial in 24 patients of both sexes aged between 30 and 60 years, with a diagnosis of metabolic syndrome according to the modified International Diabetes Federation (IDF) criteria, without treatment.

They will be assigned randomly two groups of 12 patients, each to receive 150 mg of ursolic acid or placebo before breakfast for 12 weeks.

Insulin sensitivity will be calculated by Matsuda Index with dates from glucose and insulin levels from Oral Glucose Tolerance Test; Waist circumference will be measured; triglycerides and High density lipoprotein (HDL-C) and blood pressure will be evaluated before and after intervention in both groups.

Statistical analysis will be presented through measures of central tendency and dispersion, average and deviation standard for quantitative variables; frequencies and percentages for variable qualitative. Qualitative variables will be analyzed by X2, will be used for differences inter-group Mann-Whitney U Test and Wilcoxon Test for the within-groups differences. Will be considered statistical significance p ≤0.05.

This protocol was approved by a local ethics committee (CEI/075/2014) and written informed consent will be obtained from all volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed
* Patients both sexes
* Age between 30 and 60 years
* Metabolic Syndrome according to the IDF criteria:
* Waist circumference Man ≥90 cm, Woman ≥80 cm; and two of the following criteria:
* High density lipoprotein Man ≤40 mg/dL, Woman ≤50 mg/dL;
* Fasting glucose ≥100 mg/dL;
* Triglycerides ≥150 mg/dL;
* Blood pressure ≥130/85 mmHg

Exclusion Criteria:

* Women with confirmed or suspected pregnancy
* Women under lactation and/or puerperium
* Hypersensibility to ursolic acid o calcined magnesia
* Physical impossibility for taking pills
* Known uncontrolled renal, hepatic, heart or thyroid diseased
* Previous treatment for the metabolic syndrome components
* Body Mass Index ≥39.9 kg/m2
* Fasting glucose ≥126 mg/dL
* Triglycerides ≥500 mg/dL
* Total cholesterol ≥240 mg/dL
* Low density lipoprotein (c-LDL) ≥190 mg/dL
* Blood Pressure ≥140/90 mmHg

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel González-Ortíz, PhD, Principal Investigator — University of Guadalajara
Locations (1):
- Instituto de Terapéutica Experimental y Clínica, Guadalajara, Jalisco, Mexico

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ursolic Acid | Placebo
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ursolic Acid | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (8.5) | 46.5 (8.7) | 45.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  Mexico | 12 | 12 | 24
Total Insulin Sensitivity [Mean (Standard Deviation); unit: index] — Matsuda Index value is used to indicate insulin resistance on diabetes. Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]. The entered values reflect the insulin sensitivity
  index | 3.1 (1.1) | 3.1 (0.6) | 3.1 (0.8)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 93 (9) | 97 (10) | 95 (10)
Fasting Glucose [Mean (Standard Deviation); unit: mmol/L] | 6.0 (0.5) | 5.8 (0.9) | 5.9 (0.7)
Triglycerides [Mean (Standard Deviation); unit: mmol/L] | 2.0 (0.6) | 2.5 (0.1) | 2.3 (0.4)
High Density Lipoprotein cholesterol (HDL-c) [Mean (Standard Deviation); unit: mmol/L] | 1.6 (0.6) | 1.8 (0.7) | 1.7 (0.7)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 125 (13) | 128 (20) | 127 (17)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 77 (12) | 80 (10) | 78 (11)
Body Weight [Mean (Standard Deviation); unit: kg] | 75.7 (11.5) | 81.5 (14.0) | 78.6 (12.8)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.9 (3.6) | 31.7 (4.2) | 30.8 (3.9)
Total Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 6.0 (1.4) | 6.0 (2.0) | 6.0 (1.7)
Low Density Lipoproteins cholesterol (LDL-c) [Mean (Standard Deviation); unit: mmol/L] | 3.7 (1.1) | 3.5 (2.1) | 3.6 (1.6)
Creatinine [Mean (Standard Deviation); unit: µmol/L] | 61.1 (18.6) | 68.1 (15.0) | 64.6 (16.8)
Uric acid [Mean (Standard Deviation); unit: µmol/L] | 243.9 (53.5) | 291.5 (71.4) | 267.7 (62.5)

OUTCOME MEASURES:

1. Primary Outcome: Total Insulin Sensitivity
Description: The insulin sensitivity was calculated at baseline and at week 12. The value reported corresponds at week 12 with Matsuda index. Matsuda Index value is used to indicate insulin resistance on diabetes.
  Insulin sensitivity was calculated with Matsuda index [10,000 / √glucose 0' x insulin 0') (mean glucose oral glucose tolerance test (OGTT) x mean insulin OGTT)]. The entered values reflect the insulin sensitivity
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: index
Arm/Group | Ursolic Acid | Placebo
Number analyzed (Participants) | 12 | 12
index | 4.2 (1.2) | 2.6 (1.4)
Statistical Analysis 1: Comparison: Ursolic Acid vs Placebo; Test type: Other; p = 0.003, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Waist Circumference
Description: Waist circumference was evaluated at baseline and at week 12 with a flexible tape and the entered values reflect the waist circumference measure at week 12
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Ursolic Acid | Placebo
Number analyzed (Participants) | 12 | 12
cm | 83 (9) | 96 (8)
Statistical Analysis 1: Comparison: Ursolic Acid vs Placebo; Test type: Other; p = 0.008, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Fasting Glucose
Description: The fasting glucose levels were evaluated at baseline and week 12 with enzymatic/colorimetric techniques and the entered values reflect the fasting glucose level at week 12
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ursolic Acid | Placebo
Number analyzed (Participants) | 12 | 12
mmol/L | 4.7 (0.4) | 5.7 (0.7)
Statistical Analysis 1: Comparison: Ursolic Acid vs Placebo; Test type: Other; p = 0.002, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Triglycerides
Description: The triglycerides were evaluated at baseline and week 12 with enzymatic-colorimetric techniques and the entered values reflect the triglycerides level at week 12
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ursolic Acid | Placebo
Number analyzed (Participants) | 12 | 12
mmol/L | 1.8 (0.8) | 2.5 (1.3)
Statistical Analysis 1: Comparison: Ursolic Acid vs Placebo; Test type: Other; p = 0.308, Wilcoxon (Mann-Whitney)

5. Primary Outcome: High Density Lipoprotein Cholesterol (HDL-c)
Description: The HDL-c levels were evaluated at baseline and week 12 with enzymatic/colorimetric techniques and the entered values reflect the c-HDL level at week 12
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ursolic Acid | Placebo
Number analyzed (Participants) | 12 | 12
mmol/L | 1.8 (0.9) | 1.8 (0.7)
Statistical Analysis 1: Comparison: Ursolic Acid vs Placebo; Test type: Other; p = 0.575, Wilcoxon (Mann-Whitney)

6. Primary Outcome: Systolic Blood Pressure
Description: The systolic blood pressure was evaluated at baseline and week 12 with a digital sphygmomanometer and the entered values reflect the systolic blood pressure at week 12
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ursolic Acid | Placebo
Number analyzed (Participants) | 12 | 12
mmHg | 120 (8) | 124 (15)
Statistical Analysis 1: Comparison: Ursolic Acid vs Placebo; Test type: Other; p = 0.169, Wilcoxon (Mann-Whitney)

7. Primary Outcome: Diastolic Blood Pressure
Description: The diastolic blood pressure was evaluated at baseline and week 12 with a digital sphygmomanometer and the entered values reflect the diastolic blood pressure at week 12
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Ursolic Acid | Placebo
Number analyzed (Participants) | 12 | 12
mmHg | 76 (6) | 76 (7)
Statistical Analysis 1: Comparison: Ursolic Acid vs Placebo; Test type: Other; p = 0.373, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Body Weight
Description: The body weight was measured at baseline and week 12 with a bioimpedance balance and the entered values reflect the weight at week 12
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Ursolic Acid | Placebo
Number analyzed (Participants) | 12 | 12
kg | 71 (11) | 81 (15)
Statistical Analysis 1: Comparison: Ursolic Acid vs Placebo; Test type: Other; p = 0.002, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Body Mass Index
Description: The Body Mass index was calculated at baseline and at week 12 with the Quetelet index and the entered values reflect the body mass index at week 12
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Ursolic Acid | Placebo
Number analyzed (Participants) | 12 | 12
kg/m^2 | 24.9 (1.2) | 32.1 (3.9)
Statistical Analysis 1: Comparison: Ursolic Acid vs Placebo; Test type: Other; p = 0.049, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Total Cholesterol
Description: The total cholesterol was estimated by standardized techniques at baseline and week 12 and the entered values reflect the total cholesterol level at week 12
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ursolic Acid | Placebo
Number analyzed (Participants) | 12 | 12
mmol/L | 5.2 (1.2) | 6.4 (1.9)
Statistical Analysis 1: Comparison: Ursolic Acid vs Placebo; Test type: Other; p = 0.224, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Low Density Lipoproteins Cholesterol (LDL-c)
Description: The LDL-c levels were measured at baseline and at week 12 with standardized techniques and the entered values reflect the c-LDL levels at week 12
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ursolic Acid | Placebo
Number analyzed (Participants) | 12 | 12
mmol/L | 2.8 (1.2) | 4.3 (2.3)
Statistical Analysis 1: Comparison: Ursolic Acid vs Placebo; Test type: Other; p = 0.116, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Creatinine
Description: The creatinine levels were measured at baseline and at week 12 with standardized techniques and the entered values reflect the creatinine levels at week 12
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Ursolic Acid | Placebo
Number analyzed (Participants) | 12 | 12
mmol/L | 0.06 (0.02) | 0.06 (0.02)
Statistical Analysis 1: Comparison: Ursolic Acid vs Placebo; Test type: Other; p = 0.953, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Uric Acid
Description: The uric acid levels were measured at baseline and at week 12 with standardized techniques and the entered values reflect the uric acid levels at week 12
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Ursolic Acid | Placebo
Number analyzed (Participants) | 12 | 12
µmol/L | 249.8 (53.5) | 422.3 (124.9)
Statistical Analysis 1: Comparison: Ursolic Acid; Test type: Other; p = 0.999, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Throughout the study (12 weeks)
Arm/Group | Ursolic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/12 | 6/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ursolic Acid (N=12) | Placebo (N=12)
Abdominal distention (Gastrointestinal disorders) | 3 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes